CLINICAL TRIAL: NCT01548261
Title: Donating Oral Mucosal Cells for the Study of ex Vivo Culture of Cells Sheets
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, Wei-Li Chen/Assistant Professor, National Taiwan University, Department of Ophthalmology., National Taiwan University Hospital
Other Study IDs: 201110051RB
Record Dates: First submitted 2012-03-05; First posted 2012-03-08 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Healthy
Keywords: obtain the oral mucosal tissue from healthy donors

STUDY DESIGN:
Observational Model: Case-Only
Biospecimen Retention: Samples With DNA — Donating oral mucosal cells for the study of ex vivo culture of cells sheets.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Health people.
  Interventions: Procedure: Donating oral mucosal cells

INTERVENTIONS:
Procedure: Donating oral mucosal cells — Donating oral mucosal cells

SUMMARY:
Cultivated oral mucosal epithelial sheets on amniotic membrane have been reported to have good clinical results in treating patients with ocular surface disorders in both human and animal studies. However, such technique has not been well established in this hospital. The main purpose of this study is to obtain the discarded oral mucosal tissue from healthy donors who volunteer to donate their oral mucosa from buccal area. The obtained oral mucosal tissue will be cultured under different types (co-culture with or without 3T3 cells)。Inverted light microscopy, electron microscopy and immunostaining with K3/K12, K14, Ki67, P63, connexin 43, and involucrin will be preformed to test the effects of foreskin cell line co-culture system on cell condition. The investigators plan to start the study from Jan. 1st, 2011 to Dec. 31th, 2015. Thirty patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* The age 20 to 55 year-old healthy contributor.
* does not have disease of the oral cavity.

Exclusion Criteria:

* In the past had the oral mucosa disease, wound cicatrization bad, or hemoglutination condition not good medical history. Sickness must stop using above any anti-hemoglutination medicine one week.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Health people.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2012-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, department of Ophthalmology, Taipei, Taiwan